CLINICAL TRIAL: NCT06092216
Title: Characterizing Pyoderma Gangrenosum Lesion Regression and Remission by IL-36 Receptor Targeting With Spesolimab
Brief Title: Spesolimab in Pyoderma Gangrenosum
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The funding sponsor terminated our study and will conduct a multicenter national study in its place.
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Saakshi Khattri, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-23-00611
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Pyoderma Gangrenosum
MeSH Terms: conditions — Pyoderma Gangrenosum | interventions — spesolimab

STUDY DESIGN:
Intervention Model Description: Open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Spesolimab (Experimental): 900 mg of spesolimab intravenously (IV)
  Interventions: Drug: Spesolimab

INTERVENTIONS:
Drug: Spesolimab — 900 mg of spesolimab intravenously (IV) administered every 4 weeks at Visits 2, 3, 4, 5, 6, 7, 8, 9.
  If at visit 4 dosing schedule changes to every 3 weeks, Spesolimab will be administered at Visits 2, 3, 4, 5, 6, 8, 9, 10 and 11.

SUMMARY:
The purpose of this research study is to assess the feasibility of using spesolimab in participants with moderate to severe pyoderma gangrenosum. Pyoderma gangrenosum is a rare, inflammatory, autoimmune condition which results in ulceration of skin. The study will also investigate the body's immune response to the spesolimab (when the body detects and defends itself against substances that appear unknown and harmful).

DETAILED DESCRIPTION:
To date, there is no gold standard for treatment of PG. Patients with pyoderma gangrenosum suffer from severe pain and poor quality of life due to frequent dressing changes and disfiguring lesions. More importantly, rapidly progressing ulcers present an important risk for infection, morbidity, and mortality for patients. Spesolimab is humanized antagonistic monoclonal IgG1 antibody that blocks human IL36R signalling and subsequent downstream pro-inflammatory pathways. The IL-36 receptor blocker was recently approved for generalized pustular psoriasis (GPP). The research team hypothesize that targeting IL-36 in refractory, ulcerative postoperative PG may result in regression and resolution of a patient's lesions.

There are, at minimum, a total of 14 or 15 visits which will include physical exams, blood testing and infectious disease testing, completing questionnaires, and photographs and assessment of skin affected by PG. Spesolimab will be administered via a 90-minute infusion every 3 or 4 weeks (depending on response at Visit 4) at 8 or 9 Visits during the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥ 18 years of age at the time of signing the informed consent document
* Subject is able to understand and voluntarily sign an informed consent document prior to participation in any study assessments or procedures
* Subject is able to adhere to the study visit schedule and other protocol requirements.
* Subject has clinically diagnosed ulcerative PG with PARACELSUS score greater than or equal to 10
* Subject has at least one clinically measurable ulcerative PG lesion on body that has failed to respond to at least one prior therapy such as (but not limited to) topical corticosteroids, intralesional triamcinolone, prednisone, cyclosporine, IL-23 inhibitor, IL-17 inhibitors, IL-1 inhibitors, or TNF-α- blocker therapy
* Subject has moderate to severe PG as determined by a GPG severity score of ≥3
* Subject is judged to be in otherwise good overall health as judged by the investigator, based on medical history, limited physical examination, and laboratory testing. (NOTE: The definition of good health means a subject does not have uncontrolled significant co-morbid conditions).
* Females of childbearing potential (FCBP) must have a negative pregnancy test at Screening and Baseline. While on investigational product and for at least 28 days after taking the last dose of investigational product, FCBP who engage in activity in which conception is possible must use one of the approved contraceptive options described below:

  * Option 1: Any one of the following highly effective contraceptive methods: hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation; or partner's vasectomy.
  * Or option 2: Male or female condom (latex condom or nonlatex condom NOT made out of natural [animal] membrane [for example, polyurethane]). PLUS one additional barrier method:

    * (a) diaphragm with spermicide
    * (b) cervical cap with spermicide;
    * or (c) contraceptive sponge with spermicide.

The female subject's chosen form of contraception must be effective by the time the female subject presents for her Baseline visit (for example, hormonal contraception should be initiated at least 28 days before first spesolimab infusion at Baseline).

Exclusion Criteria:

* Subject has a persistent or recurring bacterial infection requiring systemic antibiotics, or clinically significant viral or fungal or helminth parasitic infections, within 2 weeks of the Screening Visit. Any treatment of such infections must have been completed at least 2 weeks prior to the Screening Visit and no new/recurrent infections should have occurred prior to the Baseline Visit.
* Subject with current or history of positive human immunodeficiency virus (HIV), or congenital or acquired immunodeficiency (i.e. Common Variable Immunodeficiency [CVID]), hepatitis B or C, or active or untreated latent tuberculosis.
* Subject has clinically significant (as determined by the investigator) renal, hepatic, hematologic, intestinal, endocrine, pulmonary, cardiovascular, neurological, psychiatric, immunologic, or other major uncontrolled diseases that will affect the health of the subject during the study, or interfere with the interpretation of study results. Uncontrolled disease defined as hospitalization within 1 month of screening visit or determined by specialist (rheumatologist, gastroenterologist) consulted prior to study start.
* Subject has presence of acute demyelinating neuropathy
* Major surgery (according to the investigator's assessment) performed within 12 weeks prior to receiving first dose of spesolimab or planned during trial such as hip replacement, aneurysm removal, stomach ligation, or otherwise determined by investigator
* Subject has a suspected or active lymphoproliferative disorder or malignancy
* Subject was treated previously with spesolimab or another IL-36R inhibitor biologic
* Any documented active or suspected malignancy or history of malignancy within 5 years prior to screening, except appropriately treatment basal or squamous cell carcinoma of the skin or in situ carcinoma of uterine cervix.
* Subject has received a live attenuated vaccine ≤ 30 days prior to study initiation.
* History of adverse systemic or allergic reactions to any component of the study drug.
* Female subject who is pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-09-23 (Actual); Primary Completion 2025-01-14 (Actual); Study Completion 2025-01-14 (Actual)

PRIMARY OUTCOMES:
Change in Global Pyoderma Gangrenosum (GPG) Severity Score | Baseline and Week 16
  One point decrease on GPG severity score at week 16 from baseline in target lesion
  0. Completely clear; evidence of cribriform scarring, re-epithelization and possible residual hyperpigmentation. 0% ulceration apparent, lesion is dry.
  1. Almost clear; <25% of active ulceration present; > 90% granulation tissue present with mild pink, slightly elevated borders. Some evidence of re-epithelization. Minimal to no purulent drainage at presentation;
  2. Mild; <50% of active ulceration with perceptible border elevation with mild red border. Evidence of granulation tissue without any re-epithelization of skin. Few drops purulence appreciated upon examination.
  3. Moderate; <75% active ulceration with marked red, rolled borders and significant purulence. Some evidence of granulation tissue with multiple purulent drops and significant purulence on ulcer bed at presentation
  4. Severe; 100% active ulcer with violaceous, raised rolled borders. Necrotic tissue may be present.

SECONDARY OUTCOMES:
Number of participants with Complete re-epithelization of PG lesions | Up to Week 28
  Number of participants with Complete re-epithelization of PG lesions = GPG Score 0
  GPG Score 0 - Completely clear; evidence of cribriform scarring, re-epithelization and possible residual hyperpigmentation. 0% ulceration apparent and lesion is dry
Absolute Change in patient-reported Pain severity (Pain-VAS) score | Baseline and up to Week 28
  Absolute change at Week 28 from baseline in patient-reported pain severity (Pain-VAS).
  Patient Pain Visual Analogue Scale (VAS):
  Patients will be asked to report pain scores at each visit. Patients will report scores on a scale of 0 to 10.
  0 signifies no pain and 10 signifies the worst pain imaginable. Higher scores indicate increased levels of pain.
Absolute Change in Dermatology Life Quality Index (DLQI) | Baseline and up to Week 28
  Absolute Change at week 28 from baseline in DLQI.
  The DLQI is a validated questionnaire consisting of 10 questions that has been used in many randomized controlled trials in dermatology.
  Scoring of each question is as follows:
  Very much - 3 A lot - 2 A little - 1 Not at all - 0 Not relevant - 0 Question unanswered - 0
  The DLQI is calculated by summing the score of each question with total scale from 0-30. Higher score represents a quality of life that is more impaired.
  Definition of DLQI Scores 0-1 = no effect at all on patient's life 2-5 = small effect on patient's life 6-10 = moderate effect on patient's life 11-20 = very large effect on patient's life 21-30 = extremely large effect on patient's life
  A change in DLQI score of at least 4 points is considered clinically important. Such change suggests that there has actually been a meaningful change in that patient's quality of life since the previous measurement of his/her/their DLQI scores.
Recurrence of PG lesions (GPG >0) after achieving complete re-epithelialization (GPG score 0) and spesolimab cessation | Up to 16 week post-spesolimab last dose
  GPG Severity Score Scale:
  0. Completely clear; evidence of cribriform scarring, re-epithelization and possible residual hyperpigmentation. 0% ulceration apparent, lesion is dry
  1. Almost clear; <25% of active ulceration present; > 90% granulation tissue present with mild pink, slightly elevated borders. Some evidence of re-epithelization. Minimal to no purulent drainage at presentation
  2. Mild; <50% of active ulceration with perceptible border elevation with mild red border. Evidence of granulation tissue without any re-epithelization of skin. Few drops purulence appreciated upon exam.
  3. Moderate; <75% active ulceration with marked red, rolled borders and significant purulence. Some evidence of granulation tissue with multiple purulent drops and significant purulence on ulcer bed at presentation
  4. Severe; 100% active ulcer with violaceous, raised rolled borders. Necrotic tissue may be present. No evidence of granulation tissue. Extensive purulent drops on ulcer bed
Severity of the recurrence of PG lesions - Global Pyoderma Gangrenosum (GPG) Severity Score | Last dose (Week 26 or 28) up to 16 week post-spesolimab last dose
  Scale:
  0. Completely clear; evidence of cribriform scarring, re-epithelization and possible residual hyperpigmentation. 0% ulceration apparent and lesion is dry
  1. Almost clear; <25% of active ulceration present; more than 90% granulation tissue present with mild pink, slightly elevated borders. Some evidence of re-epithelization. Minimal to no purulent drainage at presentation
  2. Mild; <50% of active ulceration with perceptible border elevation with mild red border. Evidence of granulation tissue without any re-epithelization of skin. Few drops purulence appreciated upon examination.
  3. Moderate; <75% active ulceration with marked red, rolled borders and significant purulence. Some evidence of granulation tissue with multiple purulent drops and significant purulence on ulcer bed at presentation
  4. Severe; 100% active ulcer with violaceous, raised rolled borders. Necrotic tissue may be present. No evidence of granulation tissue. Extensive purulent drops present on ulcer bed

CONTACTS AND LOCATIONS:
Overall Officials: Saakshi Khattri, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Data will be analyzed as aggregated data.

DOCUMENTS (1):
  • Informed Consent Form (2024-08-06): https://cdn.clinicaltrials.gov/large-docs/16/NCT06092216/ICF_000.pdf